CLINICAL TRIAL: NCT02643212
Title: Multicenter Prospective Randomized Trial of the Effect of Rivaroxaban on Survival and Development of Complications of Portal Hypertension in Patients With Cirrhosis
Acronym: CIRROXABAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: David Garcia Cinca (Other)
Collaborators: IDIBAPS - Dr. Juan Carlos García Pagán (Unknown)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Project Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-005523-27
Record Dates: First submitted 2015-10-26; First posted 2015-12-31 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Rivaroxaban (Experimental): Rivaroxaban 10mg, 1 once a day
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban
  Arms: Rivaroxaban
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main objective of the study will determine if patients with liver cirrhosis, anticoagulation free survival improves hypertension decompensation portal and / or transplantation without serious side effects. For it is conduct a double-blind multicenter clinical trial in which patients will be randomized to receive Rivaroxaban or placebo. It included 160 patients with liver cirrhosis and insufficiency mild to moderate hepatic. It will also analyze and develop secondary endpoint portal vein thrombosis. The confirmation of our hypothesis would lead to a radical change in treatment of patients with cirrhosis include treatment with Rivaroxaban in its drove.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years of both sexes.
* Clinical and / or laboratory criteria, ultrasound and / or liver biopsy compatible with the diagnosis of viral cirrhosis (If hepatitis B virus: hepatitis B virus-DNA must be negative; if hepatitis C virus: sustained virologic response should be at least for 6 months prior to enrollment); alcohol (in the last 6 months: in men less than 60 g daily intake in women less than 40 g); nonalcoholic steatohepatitis and cryptogenic.
* Presence of clinically significant portal hypertension defined by clinical criteria (presence of esophageal varices or ascites), elastography (liver Fibroscan® ? 21 kPa) or hemodynamic (Hepatic venous pressure gradient > 10 mmHg)
* Mild to moderate hepatic impairment defined by Child-Pugh of 7-10 points.
* Written informed consent to participate in the study

Exclusion Criteria:

* Any previous or current thrombosis in splenoportal axis (must be ruled out by US-Doppler earlier than one month after randomization; if doubts: computed tomography angiography or magnetic resonance angiography if required).
* Background of hepatic encephalopathy grade II or higher
* Ascites that required prior practice of paracentesis in the last year d. Indication for use of anticoagulant and / or antiplatelet therapy for any reason.
* Hypersensitivity to the active ingredient or to excipients
* Active bleeding, clinically significant, or risk of major bleeding.
* Pregnancy and lactation.
* Hepatocellular carcinoma or malignant neoplasia at the time of inclusion.
* Any comorbidity involving a therapeutic limitation and/or a life expectancy <12 months.
* Existence of risk bleeding esophageal varices or prior variceal bleeding. They may not be included until full treatment (stable beta blockers dosage or eradication trough varices ligation).
* Pregnancy or lactation.
* Severe thrombocytopenia <40,000 platelets / dl.
* Kidney failure (creatinine clearance <15ml / min).
* Transjugular intrahepatic portosystemic shunt or portosystemic shunt carrier.
* Child-Pugh score greater than 10.
* In hepatitis C virus liver cirrhosis patients: not carrying at least six months in sustained virologic response. In hepatitis B virus liver cirrhosis patients: hepatitis B virus DNA is not negative .
* Active alcoholism (60 g / day in men and 40 in women)
* Use of potent inhibitors of cytochrome cytochrome P450 3A4 (ketoconazole, protease inhibitor antiretroviral treatment in human immunodeficiency virus patients) or cytochrome inductors (rifampicin. Phenytoin ...).
* Participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Survival free of transplant and decompensation / complications of portal hypertension. | At month 24
  Is defined as decompensation / complications of portal hypertension:
  * significant bleeding episode (defined as Baveno V) by portal hypertension (esophageal varices, gastric varices; gastropathy Portal Hypertension)
  * Hepatic encephalopathy grade II or higher.
  * decompensation of ascites: In patients without ascites decompensation be considered the onset of clinically detectable ascites and confirmed by utrasounds de novo; whereas in those with previous ascites will be considered end-point for worsening ascites if required: a) perform two or more paracentesis evacuator in the next 6 months, or b) the completion of a Transjugular intrahepatic portosystemic shunt.

SECONDARY OUTCOMES:
Cirrhosis progression disease (bleeding episode, encephalopathy, ascitis) | At month 24
  1. Bleeding episode due to portal hypertension.
  2. Hepatic encephalopathy grade II or higher.
  3. Ascitic decompensation: In patients without ascites, decompensation defined as "de novo" clinically detectable ascites; whereas in those with previous ascites is considered end-point for worsening ascites if required: a) perform two or more evacuative paracentesis in the following six months, or b) the completion of a TIPS
Development of portal vein thrombosis detected by ultrasound and confirmed by CT angiography or MRI angiography | At month 24
To evaluate the efficacy in preventing complications of portal hypertension | At month 24
  Development of complications of portal hypertension (anamnesis, physical examination, ultrasound and fibrogastroscopy)
Security of rivaroxaban in patients with liver cirrhosis, number of adverse events and adverse reactions in each arm of study. History and clinical evaluation of bleeding and monitoring of hematocrit. Evaluation of liver function | At month 24
  Evaluate number of bleeding episodes, hematocrit values and number of adverse events and reactions.
To evaluate the incidence of hepatocellular carcinoma | At month 24
  Incidence of hepatocellular carcinoma by semiannual ultrasound.
Effect on splenic and liver elasticity measured by fibroscan and / or acoustic radiation force impulse. | At month 24
  Effect of rivaroxaban on liver fibrosis assessed by liver elastography measured by fibroscan and / or acoustic radiation force impulse at baseline and every six months conditions.
Effect of Rivaroxaban on hepatocellular function estimated by the Child-Pugh and the model for end-stage liver disease scores. | At month 24
To correlate levels of anti-factor Xa and Rivaroxaban on survival free of transplant, cirrhosis progression disease (bleeding episode, encephalopathy, ascitis) and number of adverse events and reactions. | At month 24
  To correlate levels of Rivaroxaban and anti-factor Xa to the efficacy and safety of the drug. Rivaroxaban
To evaluate the effect of Rivaroxaban on hepatic venous pressure gradient | At month 24
  Effect on hepatic venous pressure gradient. Determination of hepatic venous pressure gradient at baseline and 12 months rivaroxaban or placebo
To assess if Rivaroxaban reduces concentration of intestinal fatty acid binding protein, 16S ribosomal DNA, CD14, interleukin 6, lipopolysaccharide binding protein and lipopolysaccharide | At month 24
  Assess Rivaroxaban reduces bacterial translocation and proinflammatory cytokines. Correlation with clinical events.

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital German Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau., Barcelona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Hospital Universitario Tenerife, Santa Cruz de Tenerife
  - Hospital universitari i politècnic La Fe de Valencia, Valencia

REFERENCES:
- [Derived] Puente A, Turon F, Martinez J, Fortea JI, Guerra MH, Alvarado E, Pons M, Magaz M, Llop E, Alvarez-Navascues C, Navarrete AA, Berenguer M, Masnou H, Banares R, Casado M, Ampuero J, Rios J, Saavedra C, Blasi A, Lisman T, Figuero CR, Huelin P, Tellez L, Arraez DM, Rodriguez M, Aguilera V, Arias Loste MT, Baiges A, Hernandez-Gea V, Perello C, Calleja JL, Genesca J, Villanueva C, Gonzalez-Alayon C, Albillos A, Crespo J, Garcia-Pagan JC. Rivaroxaban to prevent complications of portal hypertension in cirrhosis: The CIRROXABAN study. J Hepatol. 2025 Nov;83(5):1069-1076. doi: 10.1016/j.jhep.2025.06.035. Epub 2025 Jul 19. PMID 40691992